CLINICAL TRIAL: NCT01873898
Title: Clinical Investigation of the Rex Medical -Closer™ Vascular Closure System -Reduced Time to Ambulation Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rex Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REX-OUS-2027-004
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Bleeding
Keywords: femoral artery; access site; hemostasis
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): This is a single arm, prospective study to collect data on the safety and effectiveness of the Rex Medical Closer™ Vascular Closure System. Only subjects who are scheduled to undergo an interventional diagnostic procedure that requires closure of the femoral access site are eligible for study participation.
  Interventions: Device: Rex Medical Closer™ Vascular Closure System

INTERVENTIONS:
Device: Rex Medical Closer™ Vascular Closure System — The Rex Medical CloserTM Vascular Closure System is currently being investigated for use in closing and reducing time to hemostasis at the femoral arterial puncture site in subjects who have undergone diagnostic angiography procedures or interventional procedures using up to a 7 French procedural sheath. This study will evaluate the safety and efficacy of the Rex Medical CloserTM Vascular Closure System to close the femoral artery access site of subjects who have undergone diagnostic angiography procedures with early ambulation and discharge as soon as possible after sheath removal and device placement.
  Other Names: Closer™

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Rex Medical Closer™ Vascular Closure System to close the femoral arterial puncture site in subjects who have undergone diagnostic angiography procedures with early ambulation and discharge.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age.
* Subject is able to undergo diagnostic angiography procedure and is found suitable to receive such a device at the femoral arterial puncture site in order to reduce time to hemostasis.
* Subject or his/her legal guardian understands the nature of the procedure, and provides written informed consent prior to the procedure.
* Subject is available and willing to participate in follow-up through 30 days post femoral closure.

Exclusion Criteria:

* Subject with known allergies to polylactic acid (PLA), polyglycolic acid (PGA) or polydioxanone (PDO) polymers
* Subject with severe acute non-cardiac systemic disease
* Subject with evidence of systemic infection
* Subject where bacterial contamination of the procedural sheath or surrounding tissues may have occurred as this may increase risk of infection
* Subject with coagulopathy (bleeding disorders, including thrombocytopenia, hemophilia, etc.)
* Subject taking thrombolytic medication which reduces fibrinogen to less than 100 mg/dl
* Subject who has had a previous arterial access in the femoral artery on the treatment side with an existing hematoma >5 cm in diameter
* Subject who is unable to ambulate at baseline
* Subject who has had another closure device used in the treatment side within the previous 90 days
* Subject who requires re-entry of the treatment side planned within the next 90 days post-procedure
* Subject has a history of surgical repair on the treatment side
* Subject has planned surgeries for any reason within 90 days post- procedure
* Subject is pregnant or is lactating (non-pregnancy must be confirmed by testing)
* Has a history of a psychiatric condition, substance abuse or alcohol abuse that, in the opinion of the investigator, will potentially interfere with his or her participation
* Subject has been previously enrolled in the Rex Closer™ study
* Subject who is currently or within the previous 4 weeks been enrolled in another investigational device or drug trial
* Subject is incarcerated at the time of enrollment
* Subject where the procedural sheath has been placed through the superficial femoral artery and into the profundafemoris
* Subject where the procedure puncture site is at or distal to the bifurcation of the superficial femoral profundafemoris artery, as this may result in 1) the intravascular sealing patch catching on the bifurcation or being positioned incorrectly, and/or 2) intravascular deployment of the device into the vessel (These events may reduce blood flow through the vessel leading to symptoms of distal arterial insufficiency.)
* Subject's procedure was accessed through a vascular graft
* Subjects with uncontrolled hypertension (> 230 mm Hg systolic)
* Subjects with small femoral artery size (Less than 5 mm in diameter)
* Subjects with stenosis > 50% at the vicinity of the femoral arterial puncture site
* Subjects with anomalous branches or vessel abnormalities present in the vicinity of the femoral arterial puncture site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Time to Ambulation | Day 0
  Time to Ambulation - in minutes, defined as the time from when hemostasis is achieved to the time when ambulation is achieved (patient standing and walking at least 6.1 meters [20 feet] without re-bleeding).
Frequency of Major Adverse Events through 30 days | 30 days
  The primary safety endpoint is the frequency of Major Adverse Events through 30 days, defined as one of the following events related to the use of the investigational device: a hematoma requiring a transfusion, a device embolization, false aneurysm requiring intervention or a retroperitoneal bleed.

SECONDARY OUTCOMES:
Time to Hemostasis | Day 0
  Time to Hemostasis - in minutes, defined as the time from when the delivery system releases both sutures, which are attached to the sealing member, to the time that hemostasis (absence of expanding or developing hematoma) is achieved
Placement Technical Success | Day 0
  Placement Technical Success - defined as the successful deployment of the device at the intended placement site such that hemostasis is achieved.
Clinical Success | Day 0
  Clinical Success - evaluated from the time of device deployment, and defined as Placement Technical Success in the absence of any major safety endpoint including subsequent hematoma requiring a transfusion, a device embolization, false aneurysm requiring intervention, or retroperitoneal bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Centro de IntervencionesEndovasculares Y Cirugia Cardiovascular
Locations (1):
- Centro de IntervencionesEndovasculares Y Cirugia Cardiovascular, Asunción, Paraguay